CLINICAL TRIAL: NCT07071129
Title: Virtual Reality for Enhancement of Vision
Acronym: VR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Covid pandemic
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jeffrey L Goldberg, Principal Investigator, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 39418
Record Dates: First submitted 2025-07-09; First posted 2025-07-17 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Glaucoma; Vision Disorder
MeSH Terms: conditions — Glaucoma; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Virtual Reality Stimulation in Patients with Eye Disorders (Experimental): Participants use the VR headset for up to 1 year, followed by 1 year follow-up period.
  Interventions: Device: Virtual Reality Stimulation
- Virtual Reality Stimulation in Participants with Normal Vision (Experimental): Participants use the VR headset for up to 1 year, followed by 1 year follow-up period.
  Interventions: Device: Virtual Reality Stimulation

INTERVENTIONS:
Device: Virtual Reality Stimulation — VR 1 hour sessions will consist of an exposure to a non-invasive visual stimulation where the subject will be sitting wearing a VR headset.

SUMMARY:
This project aims to evaluate the use of Virtual Reality (VR) based visual stimulation for the treatment of blindness arising from Glaucoma and other retinal diseases or disorders of the visual system, through regeneration of axons of retinal ganglion cells (RGCs) in humans.

In certain cases of blindness, such as in Glaucoma, or in certain injuries, the optic nerves behind the retina of our eyes get damaged, leading to partial blindness, mostly near the periphery of our eye. Recent research in Dr.Huberman's laboratory has identified visual stimulation as a non-invasive model for regeneration of such damaged axons in rodents, back to the vision centers of their brain.

ELIGIBILITY:
Inclusion Criteria:

For subjects with glaucoma, other retinal diseases, or disorders of the visual system:

* 1. Patient age > 12 years
* 2. Compliance with investigator instructions, tests and visit during subject participation in the study.
* 3. Sufficient fixation ability
* 4.Best corrected visual acuity of 20/200 or better in at least one eye, or capable to see the visual stimulus at least in one eye.

For healthy volunteers:

* 1. Patient age > 12 years
* 2. Compliance with investigator instructions, tests and visit during subject participation in the study.
* 3.Best corrected visual acuity of 20/20 in both eyes.
* 4. Sufficient fixation ability

Exclusion Criteria:

* 1. Electric or electronic implants (such as cardiac pacemaker)
* 2. Any metal artifacts in the head or truncus area (with the exception of dental implants)
* 3. Epilepsy and photo-sensibility; acute auto-immune diseases
* 4. Acute conjunctivitis
* 5. Pathological nystagmus

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Goldberg, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Byers Eye Institute at Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Virtual Reality Stimulation in Patients with Eye Disorders; Virtual Reality Stimulation in Participants with Normal Vision: Participants use the VR headset for up to 2 years, followed by up to 1 year follow-up period.
Period: Overall Study
Arm/Group | Virtual Reality Stimulation in Patients with Eye Disorders | Virtual Reality Stimulation in Participants with Normal Vision
Started | 22; 32 Eyes | 0; 0 Eyes
Diagnosis of Glaucoma | 21; 31 Eyes | 0; 0 Eyes
Completed | 5; 7 Eyes | 0; 0 Eyes
Not Completed | 17; 25 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Arm/Group | Virtual Reality Stimulation in Patients With Eye Disorders
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 66.5 [16 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Field Index (VFI)
Description: VFI (expressed as a percentage) is a global measure of the visual field used to quantify the extent of visual field loss, with 100% representing a normal visual field and 0% indicating complete blindness.
Time Frame: Baseline, Month 9, Month 24
Population: Participants with data at the respective timepoint
Measure: Mean (Standard Error); unit: Percent of visual field
Units Other Than Participants: Eyes
Arm/Group | Virtual Reality Stimulation in Patients with Eye Disorders
Number analyzed (Participants) | 17
Number analyzed (Eyes) | 32
Percent of visual field
  Baseline | 55.06 (5.77)
  Month 9: number analyzed (Participants) | 10
  Month 9: number analyzed (Eyes) | 18
  Month 9 | 57.66 (6.86)
  Month 24: number analyzed (Participants) | 4
  Month 24: number analyzed (Eyes) | 5
  Month 24 | 73.5 (11.08)

2. Primary Outcome: Change in Mean Deviation Index (MD)
Description: MD is a global measure of the visual field. It is a statistical index that represents the average difference in visual field sensitivity compared to a normal age-matched population. It provides an overall measure of visual field loss in decibels, with more negative values indicating greater loss. Normal vision MD is better than -2dB, with end-stage glaucoma represented by a value of less than -20dB.
Time Frame: Baseline, Month 9, Month 24
Population: Participants with data at the respective timepoint
Measure: Mean (Standard Error); unit: Decibels
Units Other Than Participants: Eyes
Arm/Group | Virtual Reality Stimulation in Patients with Eye Disorders
Number analyzed (Participants) | 17
Number analyzed (Eyes) | 31
Decibels
  Baseline | -14.69 (1.65)
  Month 9: number analyzed (Participants) | 10
  Month 9: number analyzed (Eyes) | 18
  Month 9 | -13.33 (2.02)
  Month 24: number analyzed (Participants) | 5
  Month 24: number analyzed (Eyes) | 7
  Month 24 | -9.51 (3.17)

3. Secondary Outcome: Retinal Layer Thickness Assessed by Optical Coherence Tomography (OCT)
Description: OCT is a non-invasive imaging technique that uses light waves to create detailed, cross-sectional images of the eye, and is used to diagnose and manage various eye conditions.
Time Frame: baseline and month 9
Population: Participants with glaucoma who reliably completed treatment
Measure: Mean (Standard Error); unit: microns
Arm/Group | Virtual Reality Stimulation in Patients with Eye Disorders
Number analyzed (Participants) | 8
microns
  baseline | 70.67 (4.98)
  month 9 | 67.67 (3.18)

4. Secondary Outcome: Change in Best Corrected Visual Acuity
Description: Monocular Best Corrected Distance Visual Acuity in logMAR. Visual acuity of 20/20 = 0.00 on the logMAR scale, higher scores indicate worse vision (20/800 is the equivalent of 1.6 logMAR).
Time Frame: baseline and month 9
Population: Participants with glaucoma who reliably completed treatment
Measure: Mean (Standard Error); unit: logMAR
Arm/Group | Virtual Reality Stimulation in Patients with Eye Disorders
Number analyzed (Participants) | 8
logMAR
  Baseline | 0.34 (0.16)
  month 9 | 0.13 (0.10)

5. Other Pre Specified Outcome: Change in Pointwise Linear Regression (PLR) Index
Description: PLR is a point-specific measure of the visual field. It is a statistical method used to analyze visual field (VF) data, particularly in the context of glaucoma progression, by examining the trend of threshold sensitivity at each test location over time. It estimates the rate of change at each location, providing a detailed view of visual field deterioration.
Time Frame: baseline and 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years treatment
Arm/Group | Virtual Reality Stimulation in Patients with Eye Disorders
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Virtual Reality Stimulation in Patients with Eye Disorders (N=22)
Increased TMJ pain (Musculoskeletal and connective tissue disorders) | 1
Body Aches (Musculoskeletal and connective tissue disorders) | 1
Neurological storm (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination led to a small number of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT07071129/Prot_000.pdf